CLINICAL TRIAL: NCT03106740
Title: Imaging Glia-mediated NeuroInflammation and Treatment Efficacy (the IGNITE Study)
Brief Title: Evaluating the Role of Neuroinflammation in Low Back Pain
Acronym: IGNITE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marco Loggia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Marco Loggia, Associate Professor of Radiology and Anesthesiology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2017P000179; 1R01NS095937-01A1 (NIH)
Record Dates: First submitted 2017-03-28; First posted 2017-04-10 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain; Back Pain With Radiation; Back Pain Without Radiation; Back Pain Lower Back Chronic; Back Ache; Pain, Chronic
Keywords: Microglia; Minocycline; Magnetic Resonance Imaging; Positron Emission Tomography; Pain; Astrocytes; Glia; Human; Back Pain
MeSH Terms: conditions — Low Back Pain; Back Pain; Chronic Pain; cyclopia sequence; Pain | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minocycline Arm (Experimental): Evaluation with Magnetic Resonance-Positron Emission Tomography Imaging and/or behavioral pain assessment before and after a 2-week trial of Minocycline Hydrochloride, 100mg capsule
  Interventions: Drug: Minocycline Hydrochloride 100mg Capsule; Diagnostic Test: Magnetic Resonance-Positron Emission Tomography Imaging
- Placebo Arm (Placebo Comparator): Evaluation with Magnetic Resonance-Positron Emission Tomography Imaging and/or behavioral pain assessment before and after 2 weeks of treatment with a placebo capsule.
  Interventions: Diagnostic Test: Magnetic Resonance-Positron Emission Tomography Imaging; Other: Placebo Capsule

INTERVENTIONS:
Drug: Minocycline Hydrochloride 100mg Capsule — Minocycline 100mg will be administered by mouth daily for 2 weeks
  Other Names: Minocin; Solodyn; Dynacin; Myrac
  Arms: Minocycline Arm
Diagnostic Test: Magnetic Resonance-Positron Emission Tomography Imaging — Up to 15 millicuries of [11C]PBR28 will be administered to each subject at each imaging visit, for a maximum of 2 imaging visits.
Other: Placebo Capsule — 1 Placebo Capsule (compounded with lactose powder) will be administered by mouth daily for 2 weeks
  Arms: Placebo Arm

SUMMARY:
In this research, the study team will use brain imaging to evaluate the presence of neuroinflammation in the brains and spinal cords of patients with low back pain. The efficacy of minocycline use for low back pain treatment will also be evaluated by observing whether short-term minocycline administration will reduce neuroinflammation and low back pain symptoms.

DETAILED DESCRIPTION:
The goal of this research study is to evaluate whether the central nervous systems of those with low back pain are different from those of healthy, pain-free individuals. Specifically, the researchers will test whether "glial cells" (the immune cells of the brain and spinal cord) are more active in patients with low back pain than in healthy volunteers. The investigators' previous study showed that patients with chronic low back pain demonstrated elevations in brain levels of the 18kDa translocator protein (TSPO), a marker of glial activation.

To test this hypothesis, the study team will image the brains and spinal cords of patients suffering from low back pain using integrated magnetic resonance- positron emission tomography (MR-PET), and a radiotracer called [11C]PBR28, which tracks levels of glial activation.

The efficacy of minocycline as a treatment for chronic low back pain will also be evaluated. A recent study demonstrated a statistically significant reduction in pain in those with lumbar radiculopathy after treatment with minocycline, leading the investigators of this study to believe that minocycline may have potential efficacy in treating other back pain populations.

The study team will observe whether a short course of minocycline hydrochloride may reduce glial activation along with self-reported low back pain symptoms. To this end, patients will be evaluated clinically and/or re-scanned after completing a 2-week trial of minocycline or placebo (a sugar pill).

This study will be enrolling individuals who have been suffering from sub-acute (short-term) and chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* the ability to give written informed consent
* fluency in English
* on a stable pain treatment
* Chronic or sub-acute low back pain

Exclusion Criteria:

* no interventional pain procedures during drug trial
* contraindications to MRI and PET scanning (including presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia)
* pregnancy or breast feeding
* any use of recreational drugs in the past 6 months
* allergy to minocycline or other tetracyclines, or taking medications known to interact with minocycline
* any other contraindications to minocycline administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco L Loggia, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loggia ML, Chonde DB, Akeju O, Arabasz G, Catana C, Edwards RR, Hill E, Hsu S, Izquierdo-Garcia D, Ji RR, Riley M, Wasan AD, Zurcher NR, Albrecht DS, Vangel MG, Rosen BR, Napadow V, Hooker JM. Evidence for brain glial activation in chronic pain patients. Brain. 2015 Mar;138(Pt 3):604-15. doi: 10.1093/brain/awu377. Epub 2015 Jan 12. PMID 25582579
- [Background] Vanelderen P, Van Zundert J, Kozicz T, Puylaert M, De Vooght P, Mestrum R, Heylen R, Roubos E, Vissers K. Effect of minocycline on lumbar radicular neuropathic pain: a randomized, placebo-controlled, double-blind clinical trial with amitriptyline as a comparator. Anesthesiology. 2015 Feb;122(2):399-406. doi: 10.1097/ALN.0000000000000508. PMID 25373391
- [Derived] Mohammadian M, Morrissey EJ, Knight PC, Brusaferri L, Kim M, Efthimiou N, Murphy JP, Alshelh Z, Grmek G, Schnieders JH, Chane CA, Sandstrom A, Catana C, Gilman JM, Locascio JJ, Edwards RR, Zhang Y, Napadow V, Loggia ML. Investigating the potential of minocycline in reducing brain inflammation in chronic low back pain: a randomized, placebo-controlled mechanistic clinical trial. Pain. 2025 Apr 9;166(9):2044-2053. doi: 10.1097/j.pain.0000000000003543. PMID 40839604
- [Derived] Morrissey EJ, Alshelh Z, Knight PC, Saha A, Kim M, Torrado-Carvajal A, Zhang Y, Edwards RR, Pike C, Locascio JJ, Napadow V, Loggia ML. Assessing the potential anti-neuroinflammatory effect of minocycline in chronic low back pain: Protocol for a randomized, double-blind, placebo-controlled trial. Contemp Clin Trials. 2023 Mar;126:107087. doi: 10.1016/j.cct.2023.107087. Epub 2023 Jan 16. PMID 36657520

RESULTS

PARTICIPANT FLOW:
Groups:
- Minocycline Arm: Evaluation with Magnetic Resonance-Positron Emission Tomography Imaging and/or behavioral pain assessment before and after a 2-week trial of Minocycline Hydrochloride, 100mg capsule.
  Minocycline Hydrochloride 100mg Capsule: Minocycline administered by mouth daily for 2 weeks
  Magnetic Resonance-Positron Emission Tomography Imaging: Up to 15 millicuries of [11C]PBR28 administered to each subject at each imaging visit, for a maximum of 2 imaging visits.
- Placebo Arm: Evaluation with Magnetic Resonance-Positron Emission Tomography Imaging and/or behavioral pain assessment before and after 2 weeks of treatment with a placebo capsule.
  Placebo Capsule: Placebo (lactose powder) administered by mouth daily for 2 weeks.
  Magnetic Resonance-Positron Emission Tomography Imaging: Up to 15 millicuries of [11C]PBR28 administered to each subject at each imaging visit, for a maximum of 2 imaging visits.
Period: Overall Study
Arm/Group | Minocycline Arm | Placebo Arm
Started | 30 | 30
Completed | 25 | 23
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Partial data | 1 | 0

BASELINE CHARACTERISTICS:
Population: While 60 participants were randomized, 12 participants (5 in the minocycline arm and 7 in the placebo arm) did not complete the study, resulting in a final sample size of 48. Please see the Reasons Not Completed section of the Participant Flow table for more detailed information.
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline Arm | Placebo Arm | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.6 (16.9) | 49 (17.1) | 45.9 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 19 | 18 | 37
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48
Genotype [Count of Participants; unit: Participants] — Participants were genotyped for Ala147Thr TSPO polymorphism to predict their TSPO binding affinity for the radiotracer used in the PET scans (i.e., [11C]PBR28) and those with the Thr/Thr genotype (i.e., low-affinity binders) were excluded from further participation. Ala/Ala (i.e., GG) and Ala/Thr (i.e., GA) genotypes (high-affinity and mixed-affinity binders, respectively) were eligible for participation.
  Participants
    GG | 16 | 14 | 30
    GA | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Changes in Thalamic Standardized Uptake Value Ratio (SUVR)
Description: The ratio of the standardized uptake value (SUV; mean radioactivity divided by the injected dose by weight) of the whole thalamus divided by the SUV of the whole brain (i.e., standardized uptake value ratio or SUVR) derived from the translocator protein positron emission tomography (TSPO-PET) signal. Higher SUVR might be indicative of higher neuroinflammation.
Time Frame: The outcome measure was assessed in two time points, before and after a two-week treatment period.
Measure: Mean (Standard Deviation); unit: Standardized uptake value ratio
Arm/Group | Minocycline Arm | Placebo Arm
Number analyzed (Participants) | 25 | 23
Standardized uptake value ratio
  - Pre-treatment Thalamic SUVR | 1.188 (0.051) | 1.166 (0.056)
  - Post-treatment Thalamic SUVR | 1.189 (0.045) | 1.165 (0.054)
Statistical Analysis 1: Comparison: Minocycline Arm vs Placebo Arm; Test type: Superiority — Because relevant [11C]PBR28 PET imaging data were unavailable at the time of trial initiation to inform a power analysis of a treatment effect, we ran a power analysis of the treatment effect on the expected change in pain ratings based on a recent clinical trial using minocycline in subjects with back pain. We computed the sample size required for mixed effects between-subject and within-subject (Time: Pretest/Posttest) repeated measures ANOVA design. Alpha was set at 0.05 (two-tailed test); p = 0.956, Mixed Models Analysis — The p-value corresponds to the group-by-time interaction analysis of the primary outcome measure; Restricted maximum likelihood = 0.00, 95% CI 2-sided [-0.02 to 0.02] — Estimation parameter: Unstandardized partial regression coefficient (beta)

2. Secondary Outcome: Changes in Spinal PET Signal
Description: The standardized uptake value (SUV; mean radioactivity divided by the injected dose by weight) of the spine derived from the translocator protein positron emission tomography (TSPO-PET) signal. A higher SUV might be indicative of greater neuroinflammation.
Time Frame: 2 weeks
Reporting Status: Not Posted, anticipated posting 2027-02

3. Secondary Outcome: Rate of Change in Daily Modified Brief Pain Inventory (BPI) Severity Subscale
Description: Estimated Mean Rate of Change of BPI per Day, separately by Treatment Group (Minocycline vs. Placebo), measured as Slope of Change over Time
Time Frame: 2 weeks
Measure: Number (95% Confidence Interval); unit: The Brief Pain Inventory score per day
Arm/Group | Minocycline Arm | Placebo Arm
Number analyzed (Participants) | 25 | 23
The Brief Pain Inventory score per day | -0.04 [-0.08 to -0.026] | -0.03 [-0.062 to -0.006]

ADVERSE EVENTS:
Time Frame: Between 14 and 43 days from the pre-treatment scan.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Three types of adverse event data are to be reported: "All-Cause Mortality," "Serious," and "Other (Not Including Serious)" Adverse Events.
Arm/Group | Minocycline Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 9/30 | 15/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline Arm (N=30) | Placebo Arm (N=30)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline Arm (N=30) | Placebo Arm (N=30)
Ecchymosis (Injury, poisoning and procedural complications) | 4 (4) | 6 (6) — Bruising, pain, and swelling from the arterial line procedure.
Vasovagal syncope (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Claustrophobia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Discomfort (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) — Discomfort with study procedures (e.g., electrical stimulation, shoulder pain or dizziness from scan)
Gastrointestinal discomfort (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
COVID-19 infection (Infections and infestations) | 3 (3) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Pain after running a marathon
Skin cancer removal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03106740/Prot_SAP_000.pdf